CLINICAL TRIAL: NCT02067559
Title: Preventing Post-traumatic Stress in ICU Survivors: A Pilot Randomized Controlled Trial of ICU Diaries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Manitoba Medical Service Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H2013:460; 8-2014-07 (Other Grant/Funding Number: Manitoba Medical Services Foundation)
Record Dates: First submitted 2014-02-18; First posted 2014-02-20 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2017-05

CONDITIONS: Stress Disorders, Post Traumatic; Anxiety; Depression; Quality of Life
Keywords: Post Traumatic Stress Disorder; PTSD; Intensive Care Unit; ICU
MeSH Terms: conditions — Combat Disorders; Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- ICU Diaries (Experimental): A bound empty journal will be stored at the patient's bedside near the nurse charting area. All family members and ICU staff are invited to write in the ICU diary at any time. Instructions will be provided to the patient's family at the time of randomization and will be available at the bedside for reference. Staff instructions will be posted at charting area for staff. During the patient's stay in ICU, the diary will never leave the unit. Under no circumstances will any part of an ICU diary be duplicated. Research staff will take a photograph of the patient after consent is obtained and the photograph will be mounted on the first page of the diary. Photographs will be taken with a Polaroid camera; therefore there will be no other record of the photograph.
  Interventions: Behavioral: ICU Diary
- Psychoeducation (Experimental): The research nurse will provide a psychoeducational brochure to study participants at ICU discharge (if cognitive capacity is established) or 30 days after ICU discharge. If participants are not well enough 30 days post-discharge, they will be assessed every two weeks by research staff until the brochure is given to them. The brochure will describe procedures in the ICU (sedation, ventilation), and the delirium, hallucinations, and trauma that may result; as well as symptoms of PTSD post-ICU. It will provide instructions for follow-up, information, and emergency care. The brochure will instruct participants to contact their follow-up healthcare provider if they have any questions. The document will also be mailed to the participant's follow-up physician.
  Interventions: Behavioral: Psychoeducation
- ICU Diary plus Psychoeducation (Experimental): Participants will receive both ICU diary and psychoeducation interventions, with both documents provided at ICU-discharge, or 30 days post-discharge as above.
  Interventions: Behavioral: ICU Diary; Behavioral: Psychoeducation
- Treatment as Usual (No Intervention): No additional intervention to usual ICU care will be given.

INTERVENTIONS:
Behavioral: ICU Diary — Creation of an ICU diary: A bound empty journal will be stored at the patient's bedside near the nurse charting area. All family members and ICU staff are invited to write in the ICU diary at any time. Procedure for diary writing will follow previous research (see www.icu-diary.org).
  Arms: ICU Diaries; ICU Diary plus Psychoeducation
Behavioral: Psychoeducation — The psychoeducation brochure will describe procedures in the ICU (sedation, ventilation), and the delirium, hallucinations, and trauma that may result; as well as symptoms of PTSD post-ICU. It will provide instructions for follow-up, information, and emergency care. The brochure will instruct participants to contact their follow-up healthcare provider if they have any questions.
  Arms: ICU Diary plus Psychoeducation; Psychoeducation

SUMMARY:
The main objective of the study is to test the feasibility of the ICU diaries intervention in the ICU. The investigators do not have sufficient power to detect differences in the hypotheses below, but will use the present pilot study to inform sample size required to adequately power a follow-up randomized control trial.

(1) The investigators hypothesize that subjects exposed to a psychoeducation condition will have reduced rates of post-traumatic stress disorder (PTSD) compared to those experiencing treatment as usual (TAU). (2) The investigators hypothesize that compared to participants in the psychoeducation and TAU groups, those subjects exposed to an ICU diary, and those exposed to both ICU diary + psychoeducation conditions, will have significantly reduced rates of PTSD at follow-up. (3)The investigators hypothesize that participants exposed to the ICU diary + psychoeducation condition will have significantly lower rates of PTSD compared to those in the ICU diary alone condition.

DETAILED DESCRIPTION:
This is a randomized controlled pilot study involving patients who are in the ICU, for a minimum of 72 hrs with > 24 hrs mechanical ventilation. As is common in ICU research, proxy consent will be obtained from family members upon ICU admission. Patients will be randomized to 4 different conditions (1) treatment as usual (TAU) (2) ICU diary (3) psychoeducation (4) ICU diary + psychoeducation. The ICU diary will be created and maintained by nurses and family members for each patient randomized to condition (2) and (4), and will be given to patients by a research nurse upon discharge from the ICU. The patients in conditions (3) and (4) will receive a psychoeducational brochure detailing general treatment and sedation patients receive in the ICU, and the psychological symptoms such as depression and PTSD that can occur after a stay in the ICU. This brochure will also be sent to their follow-up physician. Patients in all conditions will be assessed at one week post-ICU for recollection of delusional memories using ICU Memory Tool (ICUMT), at one- and three-month post-ICU for baseline PTSD symptoms using Impact of Events Scale-Revised (IES-R), a commonly used measure of PTSD symptomatology, as well as measures of anxiety/depression, social support, and general health. At one and three month follow-up, the investigators will also ask patients if they had contact with their health care providers/follow-up physicians, sought mental health treatment, their general impressions of the intervention they received (diary, psychoeducation, both), and whether/how often they reviewed the document (if in conditions 2-4). The investigators will ascertain feasibility from the health care provider and family perspective by appending a short questionnaire to the diary, to be filled out each time an entry is made.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 17 years
* enrolment within 72 hours of ICU admission
* time of ICU stay is predicted to be >72 hours by ICU treatment team
* greater than 24 hours mechanical ventilation required
* understand verbal and written English

Exclusion Criteria:

* no caregiver/family available
* terminal illness with life expectancy of less than 6 months
* pre-existing cognitive impairment
* less than 24 hours of mechanical ventilation
* reason for ICU admission is suicide attempt / overdose

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2014-03; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Feasibility - enrollment of 1-2 participants per month | One year
  To test the feasibility of ICU diaries in a Canadian ICU setting by asking nurses and family members about the process of creating the diary.
  Specifically, feasibility of diary will be determined by a survey about the usability, time spent, and general comments on using the diary. Surveys will be filled by each individual making a diary entry (visitors and hospital staff).

SECONDARY OUTCOMES:
Efficacy at 90 days as determined by Impact of Event Scores (IES-R) | 90 days
  The investigators will measure patients' Impact of Event Scores - Revised (IES-R) at 90 days post-ICU discharge. These scores will be compared across the four intervention groups (ICU Diaries, Psychoeducation, ICU Diary + Psychoeducation, Treatment as Usual).
Change in IES-R 30 days post ICU discharge and access to follow up care at 90 days post ICU discharge | 30 and 90 days post ICU Discharge
  The investigators will measure differences (across treatment groups) between participant's Impact of Event Scores (IES-R) at 30 days post-discharge, and proportion of participants accessing follow-up care (psychiatric, psychological, primary care) at 90 days post-ICU discharge.
  The investigators will also assess anxiety, depression, quality of life scores, and social support scores 30 and 90 days post-ICU discharge, and measure the associations between these factors and the ICU Memory Tool (ICUMT) scores.
IES-R score of family member at 30 days post patient ICU discharge | 30 days post ICU discharge
  The investigators will assess family members of the discharged patient for IES-R scores at 30 days post-patient discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus R Blouw, MD, Principal Investigator — University of Manitoba
Locations (1):
- St. Boniface Hospital, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Davydow DS, Gifford JM, Desai SV, Needham DM, Bienvenu OJ. Posttraumatic stress disorder in general intensive care unit survivors: a systematic review. Gen Hosp Psychiatry. 2008 Sep-Oct;30(5):421-34. doi: 10.1016/j.genhosppsych.2008.05.006. Epub 2008 Jul 30. PMID 18774425
- [Background] Jones C, Backman C, Capuzzo M, Flaatten H, Rylander C, Griffiths RD. Precipitants of post-traumatic stress disorder following intensive care: a hypothesis generating study of diversity in care. Intensive Care Med. 2007 Jun;33(6):978-85. doi: 10.1007/s00134-007-0600-8. Epub 2007 Mar 24. PMID 17384929
- [Background] Backman CG, Walther SM. Use of a personal diary written on the ICU during critical illness. Intensive Care Med. 2001 Feb;27(2):426-9. doi: 10.1007/s001340000692. PMID 11396288
- [Background] Jones C, Backman C, Capuzzo M, Egerod I, Flaatten H, Granja C, Rylander C, Griffiths RD; RACHEL group. Intensive care diaries reduce new onset post traumatic stress disorder following critical illness: a randomised, controlled trial. Crit Care. 2010;14(5):R168. doi: 10.1186/cc9260. Epub 2010 Sep 15. PMID 20843344
- [Background] Jones C, Backman C, Griffiths RD. Intensive care diaries and relatives' symptoms of posttraumatic stress disorder after critical illness: a pilot study. Am J Crit Care. 2012 May;21(3):172-6. doi: 10.4037/ajcc2012569. PMID 22549573
- [Background] Cuthbertson BH, Hull A, Strachan M, Scott J. Post-traumatic stress disorder after critical illness requiring general intensive care. Intensive Care Med. 2004 Mar;30(3):450-5. doi: 10.1007/s00134-003-2004-8. Epub 2003 Sep 5. PMID 12961065
- [Derived] Kredentser MS, Blouw M, Marten N, Sareen J, Bienvenu OJ, Ryu J, Beatie BE, Logsetty S, Graff LA, Eggertson S, Sweatman S, Debroni B, Cianflone N, Arora RC, Zarychanski R, Olafson K. Preventing Posttraumatic Stress in ICU Survivors: A Single-Center Pilot Randomized Controlled Trial of ICU Diaries and Psychoeducation. Crit Care Med. 2018 Dec;46(12):1914-1922. doi: 10.1097/CCM.0000000000003367. PMID 30119073
- See also: Related Info — http://www.icu-diary.org